CLINICAL TRIAL: NCT05826275
Title: A Phase 1 Trial of TGN-S11 in Patients With Human Papillomavirus (HPV)-Associated Relapsed, Resistant or Metastatic Cancer
Brief Title: Phase 1 Trial in Patients With Human Papillomavirus (HPV)-Associated Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toragen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGN-S11
Record Dates: First submitted 2023-03-29; First posted 2023-04-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: HPV Associated Cancers
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase I, dose escalation/dose expansion study. Expansion Phase will begin in parallel one dose level lower than the highest dose deemed safe in the Dose Escalation in combination with a PD-1 checkpoint blockade.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): To determine the MTD in patients with HPV-associated cancers
  Interventions: Drug: TGN-S11
- Dose Expansion (Experimental): Dose Expansion Phase, in parallel one dose level lower than the highest dose deemed safe in Dose escalation with a PD-1 checkpoint blockade.
  Interventions: Drug: TGN-S11; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TGN-S11 — Small Molecule
Drug: Pembrolizumab — PD-1 checkpoint blockade
  Other Names: Keytruda
  Arms: Dose Expansion

SUMMARY:
This is an open-label, non-randomized, Phase I, dose escalation/dose expansion study in cohorts of patients with relapsed, resistant, or metastatic HPV-associated cancers. The Expansion Phase will begin in parallel one dose level lower than the highest dose deemed safe in the Dose Escalation in combination with a PD-1 checkpoint blockade.

ELIGIBILITY:
Inclusion Criteria:

* Prior histologically confirmed HPV-associated squamous cell carcinoma, which is relapsed, resistant, or metastatic
* Life expectancy of at least 3 months
* Dose Escalation Phase: patients who have experienced disease progression on Standard of Care Therapies

Exclusion Criteria:

* Active CNS metastases
* Have any history of seizure disorder or are taking prophylactic seizure medication
* Have an active viral, bacterial, or fungal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  To determine the maximum tolerated dose (MTD) of TGN-S11 in patients with human papillomavirus (HPV)-associated relapsed, resistant, or metastatic cancer.

SECONDARY OUTCOMES:
PK Parameters to determine the single dose | 30 days
  Cmax
Steady state pharmacokinetics (PK) of TGN-S11 | 30 days
  AUC

CONTACTS AND LOCATIONS:
Overall Officials: Neil J Clendeninn, MD, PhD, Study Director — Chief Medical Officer
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Yale University, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Company Website — https://toragen.com/